CLINICAL TRIAL: NCT04783532
Title: Feasibility and Acceptability of a Telehealth Mindfulness Intervention to Improve Outcomes of Patients With an Acute Exacerbation of Chronic Back Pain Presenting to the Emergency Department
Brief Title: Feasibility of Telehealth Mindfulness for Back Pain in the Emergency Department
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with participant enrollment and intervention engagement.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Rogelio Coronado, Research Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202543
Record Dates: First submitted 2021-02-26; First posted 2021-03-05 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Low Back Pain; Back Pain; Pain; Chronic Low-back Pain
Keywords: Mindfulness; Telehealth; Mindfulness-based intervention
MeSH Terms: conditions — Low Back Pain; Back Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth Mindfulness Program (Experimental): Telehealth mindfulness sessions
  Interventions: Behavioral: Telehealth Mindfulness Program

INTERVENTIONS:
Behavioral: Telehealth Mindfulness Program — Enrolled participants will participate in an individual (one-on-one) Telehealth-delivered (online with audio and video) mindfulness intervention with a trained mindfulness therapist. The intervention is adapted from mindfulness-based cognitive therapy and includes eight sessions lasting 75 minutes each (except the first session which lasts 90 minutes) over a 3-month period.

SUMMARY:
While guideline-directed nonpharmacological strategies for chronic low back pain are well established, optimal chronic pain management for emergency department patients has yet to be defined. Mindfulness interventions can be used for management of chronic conditions, yet are understudied as a primary approach for patients with chronic pain discharged from the emergency department. Currently, there is limited evidence examining whether an individual telehealth mindfulness intervention is a feasible and acceptable for these patients. This study will develop, pilot, and evaluate the feasibility and effects of an 8-session (12-week) telehealth mindfulness intervention for patients with an acute exacerbation of chronic low back pain

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Presenting to the emergency department to address a chief complaint of an acute exacerbation of chronic low back pain;
3. Meets NIH-supported definition of chronic low back pain (e.g., pain greater than 3 months that has resulted in pain on at least half the days in the past 6 months); and
4. English-speaking due to feasibility of utilizing a telehealth mindfulness program developed in English

Exclusion Criteria:

1. Patients requiring hospitalization for a medical severe condition or comorbidity;
2. Patients with a severe psychiatric or behavioral diagnosis or presenting symptoms, including psychosis, delirium, active suicidal ideation, or who screen positive on the Columbia Suicide Screening;
3. Patients with a history of multiple substance use or abuse;
4. Patients involved in litigation related to the chronic pain condition; and
5. Patients who are unable to comply with the telehealth intervention (i.e., unable to provide stable home address or access telehealth link on a mobile device or computer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment | 3 months after discharge from emergency department
  Proportion of eligible patients enrolled in study.
Feasibility - Retention | 3 months after discharge from the emergency department.
  Proportion of enrolled participants who complete study.
Feasibility - Session attendance | 3 months after discharge from the emergency department.
  Average number of sessions attended.

SECONDARY OUTCOMES:
Patient satisfaction with treatment | Baseline and 3 months after discharge from the emergency department.
  Single item assessing satisfaction of overall results from telehealth mindfulness program.
Patient Reported Outcomes Measurement Information System - Physical Function Short Form | Baseline and 3 months after discharge from the emergency department.
  4-item physical function short form from the 29-item Patient Reported Outcomes Measurement Information System scale. Total raw scores range from 4 to 20. A higher score indicates higher physical function, a better outcome.
Patient Reported Outcomes Measurement Information System - Pain Interference Short Form | Baseline and 3 months after discharge from the emergency department.
  4-item pain interference short form from the 29-item Patient Reported Outcomes Measurement Information System scale. Total raw scores range from 4 to 20. A lower score indicates lower pain interference, a better outcome.
Patient Reported Outcomes Measurement Information System - Pain Intensity | Baseline and 3 months after discharge from the emergency department.
  Single item from the 29-item Patient Reported Outcomes Measurement Information System scale assessing average pain intensity over the past 7 days rated on a 0 to 10 scale, with lower values indicates less pain, a better outcome.
Self-reported opioid medication use | Baseline and 3 months after discharge from the emergency department.
  Average number of pills per day (name and dose specified) and covered to morphine equivalent dose.
Self-reported return visits to the emergency department | 3 months after discharge from the emergency department.
  Single item assessing return visits to emergency department.

OTHER OUTCOMES:
Five Facet Mindfulness Questionnaire - 15 | Baseline and 3 months after discharge from the emergency department.
  15-item questionnaire assessing 5 facets of mindfulness (observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience). Facet scores range from 3 to 15. A higher score indicates higher level of mindfulness, a better outcome.
Pain Catastrophizing Scale | Baseline and 3 months after discharge from the emergency department.
  13-item questionnaire assessing thoughts and feeling when in pain. Total scores range from 0 to 52. A lower score indicates lower pain catastrophizing, a better outcome.
Pain Self-Efficacy Questionnaire | Baseline and 3 months after discharge from the emergency department.
  10-item questionnaire assessing confidence in ability to do certain things despite pain. Total scores range from 0 to 60. A higher score indicates higher pain self-efficacy, a better outcome.
Patient Reported Outcomes Measurement Information System - Depression Short Form | Baseline and 3 months after discharge from the emergency department.
  4-item depression short form from the 29-item Patient Reported Outcomes Measurement Information System scale. Total raw scores range from 4 to 20. A lower score indicates lower depression, a better outcome.
Patient Reported Outcomes Measurement Information System - Anxiety Short Form | Baseline and 3 months after discharge from the emergency department.
  4-item anxiety short form from the 29-item Patient Reported Outcomes Measurement Information System scale. Total raw scores range from 4 to 20. A lower score indicates lower anxiety, a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rogelio Coronado, PT, PhD, Principal Investigator — Vanderbilt University Medical Center; Kristin Archer, PhD, DPT, Study Director — Vanderbilt University Medical Center; Sean Collins, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States